CLINICAL TRIAL: NCT07155291
Title: Evaluation of Easy-to-Implement Intervention for Menstrual Pain in a Series of N-of-1 Trials: Study Protocol of the Menstrual Pain Intervention Among Students Study (MPIS)
Brief Title: Menstrual Pain Intervention Among Students
Acronym: MPIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Potsdam (Other)
Responsible Party: Principal Investigator, Stefan Konigorski, Dr. rer. nat., University of Potsdam
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8/2025
Record Dates: First submitted 2025-08-24; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Dysmenorrhea; Dysmenorrhea Primary; Dysmenorrhea Secondary; Dysmenorrhea Symptom
Keywords: Abdominal Self-Massage; Massage Physiotherapy; Menstrual Health; N-of-1 Trial
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Series of N-of-1 trials: The study follows an A-B-A design where A represents control/baseline periods and B represents the intervention period, with timing adjusted to individual menstrual cycle lengths.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abdominal Self-Massage (Experimental): All participants follow an ABA intervention sequence of 60 days, where A represents the control phase and B the intervention phase. The phase timing is adjusted to individual menstrual cycle lengths. During the intervention phase, participants are instructed to perform a self-administered abdominal massage. During the control phases, participants maintain usual care with no intervention. Daily symptoms are recorded throughout all phases.
  Interventions: Behavioral: Abdominal Self-Massage

INTERVENTIONS:
Behavioral: Abdominal Self-Massage — Daily self-administered visceral abdominal massage consisting of circular motions and pressure point techniques, performed for 5-20 minutes in total based on participant preference. The massage includes two parts: belly exercises (10 exercises) and pelvic exercises (3 exercises), with each exercise repeated 5-10 times or until the area feels relaxed. The app provides instructional videos and written step-by-step guides with drawings in English and German. Participants are recommended to use oil/cream, find a comfortable position, and integrate the massage into a daily routine.
  Other Names: Visceral Abdominal Self-Massage

SUMMARY:
Dysmenorrhea, or menstrual pain, is a prevalent issue among female students, which negatively influences students' productivity, academic performance, and quality of life.

This study explores a non-pharmaceutical physiotherapy method that has shown potential to decrease menstrual cramping, but research on its efficacy remains limited. The intervention is a visceral abdominal self-massage.

Because individuals tend to respond differently to physiotherapy methods, the investigators aim to assess the effect of performing the self-massage regularly on the self-reported perception of menstrual pain and related symptoms of female students in Germany, with a series of N-of-1 trials.

N-of-1 trials lasting up to 60 days are conducted with participants who regularly experience dysmenorrhea. Participants undergo a control (A) and an intervention phase (B), with a probable second control phase (A) depending on the individual cycle lengths and study start. Daily symptoms are recorded via the StudyU smartphone application. The baseline questionnaire collects demographic, lifestyle, and menstrual history information to identify potential effect modifiers. The intervention's effects will be estimated across individual and population levels. Participants will receive access to an analysis of their data.

The results may benefit individual well-being and contribute to the exploration of a more holistic approach to menstrual health.

ELIGIBILITY:
Inclusion Criteria:

* Female students living in Germany
* Have consistently experienced menstrual pain and other symptoms primarily during menstruation for at least the last three cycles
* Regular access to a smartphone on which the StudyU (https://www.studyu.health/) application can be installed
* Informed consent
* Proficiency in English or German

Exclusion Criteria:

* Age under 18 or over 45 years
* Participation in a different intervention study during the duration of this study
* Use of hormonal treatments affecting the menstrual cycle
* Confirmed or suspected pregnancy
* Presence of contraindicated disorders or diseases for massage
* Severe psychiatric conditions impairing informed consent or reliable participation
* Substance abuse (e.g., alcohol, drugs)
* Planned surgery within the next four to five months
* Doctor's advice against proceeding with the intervention

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Daily Perceived Menstrual Pain | Daily from date of enrollment until completion of individual N-of-1 trial, up to 60 days
  Participants assess the severity of menstrual pain on a visual analog scale from 0 to 10 (0=no pain, 10=worst pain imaginable).

SECONDARY OUTCOMES:
Pain Medication Intake | Daily from date of enrollment until completion of individual N-of-1 trial, up to 60 days
  Participants select which pain medication was used (if any) from a predefined list including: acetylsalicylic acid (Aspirin), butylscopolamine (Buscopan), butylscopolamine + paracetamol combinations, diclofenac (Voltaren), ibuprofen (Nurofen, Dolormin Extra), metamizole (Novalgin), naproxen (Dolormin for Women), paracetamol (Benuron), or other medications. Participants also report the number of tablets taken.
Additional Menstrual Symptoms | Daily from date of enrollment until completion of individual N-of-1 trial, up to 60 days
  Participants indicate if any of the following additional symptoms are experienced (Yes/No for each):
  * Cramps
  * Lower back pain
  * Nausea, vomiting, or diarrhea
  * Painful urination
  * Dyschezia
  * Abdominal bloating
  * Painful intercourse
  * Fatigue or difficulty concentrating
  * Fainting
  * Headaches
Mood Impact | Daily from date of enrollment until completion of individual N-of-1 trial, up to 60 days
  Participants rate how symptoms affected mood on a scale from 0 (no impact at all) to 4 (very strongly negatively).
Symptom Narrative | Daily from date of enrollment until completion of individual N-of-1 trial, up to 60 days
  Participants provide a daily free-text narrative describing their overall well-being, symptoms, and physical and emotional state.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Konigorski, Dr. rer. nat., Principal Investigator — Hasso-Plattner-Institut; Valeria Tisch, Master's Student, Principal Investigator — Hasso-Plattner-Institut

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to make anonymized data publicly available, either fully or partially, in a recognized research data repository to support further scientific research. Data obtained through the StudyU application will be published in its designated publicly available repository (https://designer.studyu.health).
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and the Statistical Analysis Plan will be made available before starting data analysis (approximately until end of November) and remain available throughout the duration of the study registration.